CLINICAL TRIAL: NCT03018470
Title: Usefulness of built-in Non-invasive Ventilator Software to Detect the Change in the Breathing Pattern of COPD Patients Under Home Mechanical Ventilation Before an Admission for Acute Exacerbation of COPD.
Brief Title: Change in Breathing Pattern on Non-invasive Ventilation of COPD Patients Under Home Mechanical Ventilation
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/015/SC
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Copd; COPD Exacerbation
Keywords: COPD; Non invasive ventilation; NIV; Acute exacerbation COPD; AECOPD; Telemonitoring
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Control cohort: Patient with COPD and home NIV admitted for planned respiratory review and without any sign of exacerbation
  Interventions: Other: Analysis of data from NIV built-in software
- Exacerbation cohort: Patient with COPD and home NIV admitted for acute exacerbation of COPD
  Interventions: Other: Analysis of data from NIV built-in software
- Outpatient exacerbation: Patient with COPD and home NIV admitted for planned respiratory review and with signs of acute exacerbation of COPD but not requiring inpatient management
  Interventions: Other: Analysis of data from NIV built-in software

INTERVENTIONS:
Other: Analysis of data from NIV built-in software — Analysis of breathing pattern using data obtained from NIV built-in software

SUMMARY:
Acute exacerbation of COPD (AECOPD) worsen prognosis and quality of life of COPD patients. Telemonitoring could be a useful tool for early identification of AECOPD. Parameters that have to be monitored are not well defined.

Patients with severe COPD may use home non-invasive ventilation (NIV). NIV have built-in software which are recording the breathing pattern of patients when used. The aim of this study is to identify ventilation parameters that are modified at the early stage of an AECOPD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed COPD according to GOLD guidelines
* Established on home non invasive ventilation for more than 2 weeks

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients admitted to Rouen Respiratory unit with established COPD and home non invasive ventilation
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-01; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change of respiratory rate at the early onset of AECOPD | 10 days

SECONDARY OUTCOMES:
Change of tidal volume at the early onset of AECOPD | 10 days
Change of leaks at the early onset of AECOPD | 10 days
Change of length of use of NIV at the early onset of AECOPD | 10 days
Change of number of breaks during the use of NIV at the early onset of AECOPD | 10 days
Change of proportion of triggered breaths during the use of NIV at the early onset of AECOPD | 10 days
Change of proportion of asynchronisms during the use of NIV at the early onset of AECOPD | 10 days
Change of the number of residual respiratory events during the use of NIV at the early onset of AECOPD | 10 days
Change of the inspiratory time during the use of NIV at the early onset of AECOPD | 10 days
Sensitivity and specificity of change in the breathing pattern under NIV to detect an AECOPD | 10 days
Correlation between the change in symptoms and in the breathing pattern under NIV | 10 days
Correlation between the length of the change in the breathing pattern under NIV and the length of inpatient stay | 10 days
Correlation between the importance of the change in the breathing pattern under NIV and the severity of the AECOPD | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Patout, MD, Principal Investigator — University Hospital, Rouen; Antoine Cuvelier, MD, PhD, Principal Investigator — University Hospital, Rouen; Sophie Blouet, Principal Investigator — University Hospital, Rouen
Locations (1):
- Service de Pneumologie, Oncologie Thoracique et Soins Intensifs Respiratoires, Rouen, Normandy, France